CLINICAL TRIAL: NCT06370169
Title: Endoscopic Ultrasound Guided Coil Embolization for Primary Prophylaxis of Gastric Varices
Brief Title: EUS Guided Coil Embolization for Primary Prophylaxis of Gastric Varices
Acronym: EUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, clinical professor, Asian Institute of Gastroenterology, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ROSC 1
Record Dates: First submitted 2023-12-21; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Gastric Varices Bleeding
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic ultrasound Placement of coil and glue (Other): Single arm study The standard treatment of bleeding gastric varices is obliteration with placement of coil and glue
  Duration 1,3,06 months for observation of gastric varices bleeding...
  Interventions: Device: Endoscopic ultrasound placement of Coil and glue

INTERVENTIONS:
Device: Endoscopic ultrasound placement of Coil and glue — The standard treatment of bleeding gastric varices is obliteration with placement of coil and glue
  Other Names: Ultrasound

SUMMARY:
The standard treatment of bleeding gastric varices is obliteration with placement of coil and glue. Our study will evaluate the efficacy of EUS guided coil as primary prophylaxis for high-risk gastric varices. All procedures will be performed with patient under deep sedation or general anaesthesia under the supervision of an anaesthesiologist.

DETAILED DESCRIPTION:
In this study Principal investigator recruiting patients with high-risk gastric varices for primary prophylaxis. Gastric varices are dilated submucosal veins in the lining of the stomach, found in patients with portal hypertension or elevated pressure in the portal venous system. The standard treatment of bleeding gastric varices is obliteration with placement of coil and glue. Our study will evaluate the efficacy of EUS guided coil as primary prophylaxis for high-risk gastric varices. All procedures will be performed with patient under deep sedation or general anaesthesia under the supervision of an anaesthesiologist. After the procedure patients will be discharged to home unless there is any indication for admission, such as significant abdominal pain, bleeding or chest pain. For enrolment into the study, patient has to sign an informed consent form which is provided at the end. First, we will do baseline evaluation of the patient which includes detailed clinical examination, routine laboratory tests, Upper GI Endoscopy, triphasic CT abdomen. The duration of study is 6 months. Only the routine tests necessary for the management of disease will be charged.

ELIGIBILITY:
Inclusion criteria: -

Each patient must meet all the following criteria to be enrolled in this study:

1. Gastric fundal varices larger than 2.0 cm in total diameter
2. High risk GV (GOV 2/IGV 1)
3. Primary prophylaxis
4. Patients with known fundal varices
5. Ability to give a signed informed consent

Exclusion criteria: -

The exclusion criteria for these volunteers will be:

1. Patients with a history of TIPS or any other portosystemic shunt procedure
2. Oesophageal stricture
3. Patient not fit for general anaesthesia
4. Secondary prophylaxis
5. Pediatric Patients (<18 years)
6. Pregnant or lactating mother
7. Not willing to participate

Ages: 18 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
The outcome will measure number of patient had achieved complete obliteration of varices | 6 months for observation
  Repeat Endoscopic ultrasound findings of residual flow

SECONDARY OUTCOMES:
Number of patient needed re intervention | 6 months for observation
  Repeat coil application on follow-up
Number of patient needed had bleeding following intervention like immediate (with in 5 days) or later (5-90 days) | 90 days
  These are the definite data which will be statistically analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Dr Ramchandani, MD DM, Study Director — Asian Institute of Gastroenterology
Locations (1):
- Asian institute of Gastroenterology, Hyderabad, Telangana, India